CLINICAL TRIAL: NCT04390321
Title: Application of Cognitive and Physical Training (LLM Care) and Related Affective Computing Systems on Persons With Special Needs (Cognitive Disorders)
Brief Title: Application of LLM Care and Related Affective Computing Systems on Persons With Special Needs
Acronym: dsLLM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aristotle University Of Thessaloniki (Other)
Responsible Party: Principal Investigator, Panos Bamidis, Assistant Professor, Aristotle University Of Thessaloniki
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 488
Record Dates: First submitted 2020-05-12; First posted 2020-05-15 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-05

CONDITIONS: Down Syndrome
Keywords: Down Syndrome; Physical training; Cognitive training; EEG
MeSH Terms: conditions — Down Syndrome

STUDY DESIGN:
Intervention Model Description: Participants are assigned to a single group following the same intervention
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Down Syndrome LLMcare (Experimental): Individuals with Down Syndrome which are able to execute the LLMcare physical and cognitive training intervention
  Interventions: Other: LLMcare

INTERVENTIONS:
Other: LLMcare — Participants will undergo 20 sessions of computerized cognitive and physical training, during a 2 month period. Both components have a duration of 30 minutes and are consecutive, but their sequence is pseudo-randomized. All sessions are conducted under supervision. Cognitive training uses the greek adaptation of the BrainHQ software (Posit Science Corporation), utilizing audiovisual stimuli, and targets memory, attention, cognitive-processing speed, orientation and social skills. Physical training is based on the WebFitForAll protocol and uses the motion sensor device Kinect. It consists of warm-up, aerobic, flexibility, strength, balance and cool down exercises.

SUMMARY:
Down syndrome (DS) is a genetic disorder characterized by specific physical characteristics (muscle degeneration) and cognitive phenotype (neurodegeneration caused by gene-overexpression that has affected memory, language, and other executive functions). DS is the most prevalent reason for intellectual impairment but is also often accompanied by other medical conditions such as Alzheimer's disease. Given the increased cognitive decline inherent to DS, especially in the later years, the development of a non-invasive intervention protocol to counterbalance this prevalence is imperative.

This study is an adaptation of the Long Lasting Memories (LLM) (NCT02267499) and the subsequent LLM Care (NCT02313935) projects, specifically tailored to meet the needs and capacity of people with DS. The study aims to examine the effectiveness and any potential benefits of cognitive and physical training, as offered via the ICT-based (non-pharmacological) intervention of LLM Care, on people with DS. It is worth investigating whether this intervention can aid the development of independent living skills in DS individuals and the possibility of counterbalancing the degeneration, both physical and cognitive, caused by the expression of the extra genes. To evaluate any physical, cognitive, behavioral, and neuroplastic benefits/effects and measure the influence (affective status of participant) of the training, the study utilizes psycho-somatometric assessments and neuroscientific (electroencephalographic, EEG-related) indices, as well as affective computing systems.

DETAILED DESCRIPTION:
Down Syndrome (DS) is a genetic disorder most commonly attributed to the trisomy of chromosome 21. It is considered the most prevalent reason for intellectual impairment. The extra chromosomic copy results in gene over-expression, which in turn is responsible for the characteristic non-uniform degeneration, affecting both cognition, and physical condition. The disorder has been linked to many underlying conditions such as early aging and Alzheimer's disease. Considering the cognitive decline that accompanies the increase in age, there is a need to develop non-invasive, counterbalancing interventions that will provide these individuals with a better quality of life and support them in acquiring and improving their skill set.

The target population is individuals with DS. The participants followed similar training schemes of the intervention, two days per week for one hour, for 10 weeks (aiming at 20 sessions/ participant), for one hour (30 minutes of cognitive and 30 minutes of physical training). Specifically, the participants completed the LLMcare protocol (combined cognitive and physical training) while a subgroup underwent measurements two times, one month apart, before initiating the intervention to serve as control.

The intervention is a based on LLM Care (NCT02313935) Integrated Healthcare System (https://www.llmcare.gr/en/home/) which is a successful example of commercializing the LLM (NCT02267499) research program (http://www.longlastingmemories.eu/), and has been customized to meet the needs and capacity of people with DS. The LLM Care (non-pharmaceutical) intervention is an integrated training system that targets nondemented and demented aging population and adopts an approach of cognitive and physical training to improve the quality of life and prolong the functionality of the elders.The main goal of this study is to quantify the effects of implementing the LLM Care intervention on people with DS, and particularly its effect on their physical status, cognition, behavior, and brain function. The study can potentially evaluate if adopting a cognitively and physically stimulating lifestyle can support DS individuals in acquiring and improving their skill set and act as and effective treatment against the physical and cognitive degeneration that is inherent to this syndrome The individuals with DS were evaluated via a battery of clinical and neuropsychological tests, and EEG measures at baseline (pre), exit (post) and one month after the training (follow up). Additionally, the training platform utilizes affective computing systems to evaluate the affective status of all participants throughout the training, and to establish a pleasant learning environment for all participants.

ELIGIBILITY:
Inclusion Criteria:

* Down syndrome individuals

Exclusion Criteria:

* Ability to execute the physical training protocol
* Ability to execute the cognitive training protocol

Ages: 5 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 46 (Actual)
Dates: Start 2017-02-22 (Actual); Primary Completion 2022-01-01 (Actual); Study Completion 2022-01-01 (Actual)

PRIMARY OUTCOMES:
Cognitive capacity (functional) | 2 months
  Change in cognitive functions as measured via the battery test WISC-III.
Physical capacity (general) | 2 months
  Change in physical function as measured via the Short Physical Performance Battery (SPPB, scale from 0 to 12)

SECONDARY OUTCOMES:
Cognitive capacity (verbal and non-verbal) | 2 months
  Change in verbal and non-verbal mental capabilities, as measured via the Ravens test.
Cognitive capacity (emotion identification) | 2 months
  Change in emotion identification as measured via the "Reading the mind in the eye" test
Physical capacity (mobility) | 2 months
  Change in functional mobility, gait and vestibular function as measured via the 10 Meter Walk test (timed score).
Physical capacity (flexibility) | 2 months
  Change in flexibility (especially in the lower back) as measured via the Sit and Reach test.
Physical capacity (upper body strength) | 2 months
  Change in upper body strength and endurance as measured via the Arm Curl test.
Physical capacity (balance) | 2 months
  Change in static balance as measured via the Stork Balance test (each leg, timed test).
Physical capacity (stability) | 2 months
  Change in dynamic stability as measured by the Four Square Step Test (FSST).
Physical capacity (mobility and balance) | 2 months
  Change in mobility, static and dynamic balance as measured via the Timed Up and Go test (timed test).
Change in current density strength of the cortical activity as measured via EEG | 2 months
  Changes in cortical activity strength caused via the training. Change is defined as statistical significance in the t-test comparison of the current density strength as reconstructed via Low Resolution Electromagnetic Tomography (LORETA) algorithm on the basis of high density EEG recordings, before compared to after the training
Change in cortical connectivity as measured via EEG | 2 months
  Changes in cortical connectivity caused via the training. Change is defined as statistical significance in the t-test comparison of the Transfer Entropy estimated from the cortical activity, as reconstructed via LORETA algorithm on the basis of high density EEG recordings, before compared to after the training.

CONTACTS AND LOCATIONS:
Locations (1):
- Laboratory of Medical Physics, AUTH, Thessaloniki, Greece

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Savvidis TP, Konstantinidis EI, Dias SB, Diniz JA, Hadjileontiadis LJ, Bamidis PD. Exergames for Parkinson's Disease Patients: How Participatory Design Led to Technology Adaptation. Stud Health Technol Inform. 2018;251:78-81. PMID 29968606
- [Background] Konstantinidis EI, Bamparopoulos G, Bamidis PD. Moving Real Exergaming Engines on the Web: The webFitForAll Case Study in an Active and Healthy Ageing Living Lab Environment. IEEE J Biomed Health Inform. 2017 May;21(3):859-866. doi: 10.1109/JBHI.2016.2559787. Epub 2016 Apr 27. PMID 28113566
- [Background] Styliadis C, Kartsidis P, Paraskevopoulos E, Ioannides AA, Bamidis PD. Neuroplastic effects of combined computerized physical and cognitive training in elderly individuals at risk for dementia: an eLORETA controlled study on resting states. Neural Plast. 2015;2015:172192. doi: 10.1155/2015/172192. Epub 2015 Apr 7. PMID 25945260
- [Derived] Anagnostopoulou A, Styliadis C, Kartsidis P, Romanopoulou E, Zilidou V, Karali C, Karagianni M, Klados M, Paraskevopoulos E, Bamidis PD. Computerized physical and cognitive training improves the functional architecture of the brain in adults with Down syndrome: A network science EEG study. Netw Neurosci. 2021 Mar 1;5(1):274-294. doi: 10.1162/netn_a_00177. eCollection 2021. PMID 33688615
- See also: Related Info — http://www.llmcare.gr